CLINICAL TRIAL: NCT04722263
Title: Primary Radiotherapy for the Treatment of Keloids: A Pilot Study
Brief Title: Radiotherapy for Keloids
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-11620; NCT04853433 (obsolete NCT alias)
Record Dates: First submitted 2021-01-08; First posted 2021-01-25 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Radiotherapy for patients with nonresectable keloids (Experimental): Patients will be seen by a treating radiation oncologist and treatment with the assigned dose schedule will be planned using either EBRT with electrons or high dose-rate radiotherapy (HDR) brachytherapy as deemed appropriate by the treating radiation oncologist. The treatment dose of 25 Gy in 5 fractions will be prescribed to the 90% isodose line.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — 25 Gy in 5 fractions
  Other Names: Radiation therapy

SUMMARY:
The purpose of this pilot study is to evaluate the safety and efficacy of radiation therapy (RT) in the treatment of unresected keloids.

DETAILED DESCRIPTION:
This will be a single-institution pilot study to evaluate the safety and efficacy of radiation therapy (RT) for the treatment of unresected keloids.

Primary Objective:

Evaluate feasibility and safety of radiation therapy only for the treatment of unresected keloids.

Secondary Objectives:

* To evaluate toxicity of RT for the treatment of unresected keloids.
* To evaluate response of keloids, either stability or decrease in size, after primary RT.
* To evaluate symptomatic response of unresected keloids to primary RT.
* To assess the effect on quality of life of primary RT for unresected keloids

After review of the literature on the use of RT for the treatment of keloids, both resected and unresected, as well as input of expert opinion and clinical experience by the study's radiation oncologists, the RT prescription dose for this study was selected to be 15 Gy, which will be divided into 5 Gy fractions delivered daily over on 3 consecutive days.

Patients will receive RT using external beam radiotherapy (EBRT), delivered via either electrons or megavoltage photons, or brachytherapy; RT modality will be based on the judgment of the treating radiation oncologist. The investigator team estimates that 15-20 patients will be able to be recruited. In successive intervals of enrollment and treatment of 5 patients (i.e., after 5, 10, and 15 patients have been enrolled), the study team will meet and perform interim analysis to evaluate the safety and efficacy of treatment. Investigators will discuss rates of toxicity and symptom management observed up to that point and determine if the study dose or protocol needs to be altered.

Patients will be evaluated frequently for treatment-related toxicities using CTCAE v5.0 up to 1 year after completion of RT. Any adverse event will be considered by the study investigators to evaluate the safety of the protocol and to determine whether changes to the dosing regimen are required.

Once patients have been identified as having a keloid that will not be surgically resected they will be referred to the radiation oncology department at Montefiore Medical Center. Patients will be seen by a treating radiation oncologist and treatment with the assigned dose schedule will be planned using either EBRT with electrons or high dose-rate radiotherapy (HDR) brachytherapy as deemed appropriate by the treating radiation oncologist.

Amendment for increased dose (3/2023): The treatment dose of 25 Gy in 5 fractions will be prescribed to the 90% isodose line. Treatments will be given on consecutive days (Monday through Friday not including weekends), and all efforts will be made to not introduce a weekend break if at between treatment fractions.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed keloid
* Surgical excision of keloid is either contraindicated or patient has declined treatment with surgical excision (Note: patients with keloids that recurred after previous resection are eligible, as long as the current keloid is either unresectable or patient has declined resection)
* Age ≥ 18
* Study specific informed consent provided

Exclusion Criteria:

* Prior RT to the area of interest that would result in overlap of radiation therapy fields
* Females of child bearing age without a negative serum pregnancy test prior to initiation of RT or unwilling to use contraception prior to and during the radiation course
* Keloids in areas where radiation therapy introduces unacceptable high risk of toxicity as determined by the treating radiation oncologist
* Uncontrolled intercurrent illness (e.g. symptomatic congestive heart failure, uncontrolled cardiac arrhythmia, or psychiatric situation) that would limit compliance with study requirements as judged by the treatment physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Treatment-related toxicities | Up to 1 year (+/- 1 month) post radiotherapy
  The number of patients with treatment related toxicities will be determined by the incidence of grade 2 or higher skin-related adverse events based on CTCAE V5.0 criteria during prescheduled study visits. The number of patients with treatment related toxicities will be reported in aggregate for all visits.

SECONDARY OUTCOMES:
Cessation of growth or shrinkage of keloids | Week 0, during treatment (as close to the end of the radiotherapy course as practicable
  The number of patients demonstrating cessation of growth or shrinkage of keloids as compared to baseline will be determined by measurements of the three dimensions of the keloid (maximum length, width, and height off the skin) during prescheduled study visits.
Cessation of growth or shrinkage of keloids | Up to 2 weeks (+/- 1 week) post radiotherapy
  The number of patients demonstrating cessation of growth or shrinkage of keloids as compared to baseline will be determined by measurements of the three dimensions of the keloid (maximum length, width, and height off the skin) during prescheduled study visits.
Cessation of growth or shrinkage of keloids | Up to 6 weeks (+/- 1 week) post radiotherapy
  The number of patients demonstrating cessation of growth or shrinkage of keloids as compared to baseline will be determined by measurements of the three dimensions of the keloid (maximum length, width, and height off the skin) during prescheduled study visits.
Cessation of growth or shrinkage of keloids | Up to 10 weeks (+/- 1 week) post radiotherapy
  The number of patients demonstrating cessation of growth or shrinkage of keloids as compared to baseline will be determined by measurements of the three dimensions of the keloid (maximum length, width, and height off the skin) during prescheduled study visits.
Cessation of growth or shrinkage of keloids | Up to 6 months (+/- 1 month) post radiotherapy
  The number of patients demonstrating cessation of growth or shrinkage of keloids as compared to baseline will be determined by measurements of the three dimensions of the keloid (maximum length, width, and height off the skin) during prescheduled study visits.
Cessation of growth or shrinkage of keloids | Up to 1 year (+/- 1 month) post radiotherapy
  The number of patients demonstrating cessation of growth or shrinkage of keloids as compared to baseline will be determined by measurements of the three dimensions of the keloid (maximum length, width, and height off the skin) during prescheduled study visits.
Quality of Life as determined by SKINDEX-16 questionnaire | During treatment. Assessed as close to the end of the radiotherapy course as practicable, up to ~1 week
  Patient quality of life will be evaluated by responses to a SKINDEX-16 questionnaire. The SKINDEX-16 questionnaire consists of 16 quality of life related questions which score patient responses on a 7-point Likert scale from 0 to 6 where 0 equates to "never bothered" and 6 equates to "always bothered" yielding an overall possible scoring range from 0-96. Lower SKINDEX-16 scores correlate to increased quality of life. Cumulative scores will be summarized and reported using means and standard deviations.
Quality of Life as determined by SKINDEX-16 questionnaire | Up to 10 weeks (+/- 1 week) post radiotherapy
  Patient quality of life will be evaluated by responses to a SKINDEX-16 questionnaire. The SKINDEX-16 questionnaire consists of 16 quality of life related questions which score patient responses on a 7-point Likert scale from 0 to 6 where 0 equates to "never bothered" and 6 equates to "always bothered" yielding an overall possible scoring range from 0-96. Lower SKINDEX-16 scores correlate to increased quality of life. Cumulative scores will be summarized and reported using means and standard deviations.
Quality of Life as determined by SKINDEX-16 questionnaire | Up to 6 months (+/- 1 month) post radiotherapy
  Patient quality of life will be evaluated by responses to a SKINDEX-16 questionnaire. The SKINDEX-16 questionnaire consists of 16 quality of life related questions which score patient responses on a 7-point Likert scale from 0 to 6 where 0 equates to "never bothered" and 6 equates to "always bothered" yielding an overall possible scoring range from 0-96. Lower SKINDEX-16 scores correlate to increased quality of life. Cumulative scores will be summarized and reported using means and standard deviations.
Quality of Life as determined by SKINDEX-16 questionnaire | Up to 1 year (+/- 1 month) post radiotherapy
  Patient quality of life will be evaluated by responses to a SKINDEX-16 questionnaire. The SKINDEX-16 questionnaire consists of 16 quality of life related questions which score patient responses on a 7-point Likert scale from 0 to 6 where 0 equates to "never bothered" and 6 equates to "always bothered" yielding an overall possible scoring range from 0-96. Lower SKINDEX-16 scores correlate to increased quality of life. Cumulative scores will be summarized and reported using means and standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Keyur J Mehta, MD, Principal Investigator — Montefiore
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guix B, Henriquez I, Andres A, Finestres F, Tello JI, Martinez A. Treatment of keloids by high-dose-rate brachytherapy: A seven-year study. Int J Radiat Oncol Biol Phys. 2001 May 1;50(1):167-72. doi: 10.1016/s0360-3016(00)01563-7. PMID 11316560
- [Background] Mankowski P, Kanevsky J, Tomlinson J, Dyachenko A, Luc M. Optimizing Radiotherapy for Keloids: A Meta-Analysis Systematic Review Comparing Recurrence Rates Between Different Radiation Modalities. Ann Plast Surg. 2017 Apr;78(4):403-411. doi: 10.1097/SAP.0000000000000989. PMID 28177974
- [Background] Borok TL, Bray M, Sinclair I, Plafker J, LaBirth L, Rollins C. Role of ionizing irradiation for 393 keloids. Int J Radiat Oncol Biol Phys. 1988 Oct;15(4):865-70. doi: 10.1016/0360-3016(88)90119-8. PMID 3182326
- [Background] Bijlard E, Timman R, Verduijn GM, Niessen FB, Hovius SER, Mureau MAM. Intralesional cryotherapy versus excision with corticosteroid injections or brachytherapy for keloid treatment: Randomised controlled trials. J Plast Reconstr Aesthet Surg. 2018 Jun;71(6):847-856. doi: 10.1016/j.bjps.2018.01.033. Epub 2018 Feb 6. PMID 29426811
- [Background] Cheraghi N, Cognetta A Jr, Goldberg D. RADIATION THERAPY for the Adjunctive Treatment of Surgically Excised Keloids: A Review. J Clin Aesthet Dermatol. 2017 Aug;10(8):12-15. Epub 2017 Aug 1. PMID 28979658
- [Background] Renz P, Hasan S, Gresswell S, Hajjar RT, Trombetta M, Fontanesi J. Dose Effect in Adjuvant Radiation Therapy for the Treatment of Resected Keloids. Int J Radiat Oncol Biol Phys. 2018 Sep 1;102(1):149-154. doi: 10.1016/j.ijrobp.2018.05.027. Epub 2018 May 17. PMID 29970316
- [Background] Goutos I, Ogawa R. Brachytherapy in the adjuvant management of keloid scars: literature review. Scars Burn Heal. 2017 Nov 10;3:2059513117735483. doi: 10.1177/2059513117735483. eCollection 2017 Jan-Dec. PMID 29799578
- [Background] Rossi AM, Nehal KS, Lee EH. Radiation-induced Breast Telangiectasias Treated with the Pulsed Dye Laser. J Clin Aesthet Dermatol. 2014 Dec;7(12):34-7. PMID 25584136
- [Background] Malaker K, Vijayraghavan K, Hodson I, Al Yafi T. Retrospective analysis of treatment of unresectable keloids with primary radiation over 25 years. Clin Oncol (R Coll Radiol). 2004 Jun;16(4):290-8. doi: 10.1016/j.clon.2004.03.005. PMID 15214654
- [Background] Kim J, Lee SH. Therapeutic results and safety of postoperative radiotherapy for keloid after repeated Cesarean section in immediate postpartum period. Radiat Oncol J. 2012 Jun;30(2):49-52. doi: 10.3857/roj.2012.30.2.49. Epub 2012 Jun 30. PMID 22984682
- [Background] Lo TC, Seckel BR, Salzman FA, Wright KA. Single-dose electron beam irradiation in treatment and prevention of keloids and hypertrophic scars. Radiother Oncol. 1990 Nov;19(3):267-72. doi: 10.1016/0167-8140(90)90153-n. PMID 2126387
- [Background] Chren MM, Lasek RJ, Sahay AP, Sands LP. Measurement properties of Skindex-16: a brief quality-of-life measure for patients with skin diseases. J Cutan Med Surg. 2001 Mar-Apr;5(2):105-10. doi: 10.1007/BF02737863. Epub 2001 Mar 21. PMID 11443481